CLINICAL TRIAL: NCT05833958
Title: Polypill Versus Metformin in New Onset Type 2 Diabetes: a Low Dose Triple Therapy Polypill Versus Metformin for Glycaemic Control in Newly Diagnosed Type 2 Diabetes
Brief Title: Polypill Versus Metformin in New Onset Type 2 Diabetes
Acronym: PiVOT
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The sponsor has determined that this study will be postponed due to changing business priorities.
Sponsor: George Medicines PTY Limited (Industry)
Collaborators: Brandon Biocatalyst (Unknown); The George Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GMRx-4 IR
Record Dates: First submitted 2023-03-31; First posted 2023-04-27 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GMRx-4 IR polypill in the morning and metformin Immediate Release (IR)175mg at night (Experimental): One GMRx-4 IR polypill capsule (metformin IR 175mg + dapagliflozin 2.5mg + sitagliptin 17.5mg) in the morning and one metformin IR 175mg capsule at night. Capsules are taken with, or just after, food, and swallowed whole with water. Capsules will be taken at, or as close as possible to, the same time of morning (GMRx-4 IR) and the same time of evening (metformin 175mg) each day for 16 weeks.
  Interventions: Drug: GMRx-4 IR polypill - sitagliptin, dapagliflozin, metformin; Drug: Metformin
- Metformin IR 500mg in the morning and at night (Active Comparator): One metformin IR 500mg capsule in the morning and at night. Capsules are taken with, or just after, food, and swallowed whole with water. Capsules will be taken at, or as close as possible to, the same time of morning and the same time of evening each day for 16 weeks.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: GMRx-4 IR polypill - sitagliptin, dapagliflozin, metformin — As described previously
  Arms: GMRx-4 IR polypill in the morning and metformin Immediate Release (IR)175mg at night
Drug: Metformin — As described previously - Experimental Arm, 175mg at night
  Arms: GMRx-4 IR polypill in the morning and metformin Immediate Release (IR)175mg at night
Drug: Metformin — As described previously - Active Comparator Arm, 500mg in the morning and 500mg at night
  Arms: Metformin IR 500mg in the morning and at night

SUMMARY:
The goal of this clinical trial is to learn about the effect of the GMRx-4 IR polypill compared to metformin monotherapy on glycosylated haemoglobin (HbA1c) when used as first line therapy in adults with recently diagnosed Type 2 Diabetes. The main question it aims to answer is:

That the GMRx-4 IR polypill, compared to metformin, will improve glucose lowering in those with recently diagnosed Type 2 Diabetes.

Participants will be required to take either:

One capsule of the GMRx-4 IR polypill each morning and one 175mg metformin capsule each evening for 16 weeks.

Or One metformin 500mg capsule each morning and each evening for 16 weeks.

Participants will not know which of the two treatment regimens they will be taking. Participants will be provided with the necessary guidance information, equipment, online support and telephone/video calls from trained members of the study team to complete the study procedures at home although some support from a Healthcare Professional either at home or at a clinic will be offered if needed. The study will involve participants completing the following information and procedures and reporting electronically:

Medical History (conditions and treatments) Gender Age Ethnicity/Race Weight Height Blood Pressure Heart Rate Blood collection for measurement of HbA1c (average blood glucose levels over a period of time), fasting glucose, creatinine and estimated glomerular filtration rate (eGFR) for kidney function, cholesterol, pregnancy (if not measured in a urine sample) Urine pregnancy test in women of child-bearing potential Concomitant Medications taken Safety outcomes Tolerability to the study treatment Adherence with taking the study treatment The number of any unused study treatment capsules

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years;
2. Diagnosis of Type 2 Diabetes (T2D) within 24 months;
3. Drug naïve or using metformin monotherapy at ≤1g daily;
4. Body mass index between 18.5 and 45 kg/m2;
5. HbA1c ≥6.0% (metformin monotherapy) or ≥6.5% (drug naïve), and ≤12%;
6. eGFR ≥45 ml/min/1.73m2;
7. Signed informed consent; and
8. Willingness to take a pregnancy test prior to starting treatment (participants of childbearing potential).

Exclusion Criteria:

1. There is a definite contraindication to either metformin, SGLT2 inhibitors or Dipeptidyl-peptidase 4 (DPP4) inhibitors;
2. There is a definite indication for an SGLT2 inhibitor;
3. A known situation where medication might be altered for a significant length of time (e.g., planned surgery);
4. Moderate or severe anaemia (Hb< 100g/L women and <110g/L in men), haemolytic anaemia or known haemoglobinopathy (which may affect the accurate measurement of HbA1c);
5. Unlikely to complete the trial, adhere to the trial or complete study contacts, including at-home pathology tests, according to investigator judgement; or
6. Known or suspected pregnancy or breast-feeding;
7. Participants of childbearing potential (participants who are anatomically and physiologically capable of becoming pregnant), or have a partner of childbearing potential, not willing to use highly effective contraceptive for the 16-week duration of the trial, and who do not confirm a negative pregnancy test before starting the drug;
8. Any severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgement of the Investigator, and in discussion with the Medical Monitor, would make the participant inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Change in glycosylated haemoglobin (HbA1c) | 16 weeks
  Change in glycosylated haemoglobin (HbA1c) from baseline to 16 weeks

SECONDARY OUTCOMES:
Change in fasting plasma glucose | 16 weeks
  Change in fasting plasma glucose from baseline to 16 weeks
Change in cholesterol | 16 weeks
  Change in fasting total cholesterol, LDL-cholesterol and HDL-cholesterol from baseline to 16 weeks
Change in triglycerides | 16 weeks
  Change in fasting triglycerides from baseline to 16 weeks
Change in blood pressure | 16 weeks
  Change in systolic and diastolic blood pressure from baseline to 16 weeks
Change in weight in kilograms | 16 weeks
  Change in weight from baseline to 16 weeks
Medication adherence | 16 weeks
  Medication adherence throughout the trial. Adherence will be assessed by self-report surveys entered directly into the ePRO platform (eCRF).
Medication tolerability | 16 weeks
  Medication tolerability throughout the trial (based on permanent drug cessation due to side effects and incidence of reported side effects). Tolerability will be assessed by recording of adverse effects into self-report surveys, and adverse events identified by the Investigator during study contacts, entered directly into the ePRO platform (eCRF).

IPD SHARING:
Plan to Share IPD: No
If the sponsor receives a request for study-level data listing, then such requests will be reviewed by a committee that is composed of sponsor representation and steering committee members.